CLINICAL TRIAL: NCT01256229
Title: OUTCOMES IN CHILDREN WITH DEVELOPMENTAL DELAY AND DEAFNESS: A PROSPECTIVE, RANDOMIZED TRIAL
Brief Title: Outcomes In Children With Developmental Delay And Deafness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, John S. Oghalai, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DC010075 (NIH); R01DC010075 (NIH); eProtocol #19249
Record Dates: First submitted 2010-11-12; First posted 2010-12-08 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Deafness; Hearing Loss
Keywords: deafness; hearing loss; developmental delay; mental retardation
MeSH Terms: conditions — Deafness; Hearing Loss; Learning Disabilities; Intellectual Disability | interventions — Cochlear Implantation; Hearing Aids

ARMS (3):
- Developmentally delayed - Hearing aids (Experimental): This arm contains deaf children that have developmental delays and are randomized to be treated with the conventional therapy, hearing aids.
  Interventions: Device: hearing aids
- Developmentally Delayed - Cochlear implant (Experimental): This arm contains deaf children that have developmental delays and are randomized to be treated with cochlear implantation.
  Interventions: Device: cochlear implantation
- Not developmentally delayed (Active Comparator): This control arm contains deaf children that do not have developmental delays and will be treated with cochlear implantation.
  Interventions: Device: cochlear implantation

INTERVENTIONS:
Device: cochlear implantation — This is the experimental therapy for deaf children with developmental delays, and the conventional therapy for deaf children without developmental delays.
  Arms: Developmentally Delayed - Cochlear implant; Not developmentally delayed
Device: hearing aids — This is the conventional therapy for deaf children with developmental delays.
  Arms: Developmentally delayed - Hearing aids

SUMMARY:
Children with special needs require complex, individualized therapy to maximize their long-term quality of life. One subset of children with special needs includes those with both developmental delays and deafness. Currently, there is little compelling evidence supporting the idea that cochlear implantation provides benefit to children that don't have the cognitive potential to develop normal speech and language.

We will perform a prospective, randomized clinical trial to answer the question of which intervention provides more benefit to this population of children using validated, norm-referenced tests.

Our long-term goal is to develop guidelines that may help when selecting a treatment for hearing loss in a child with developmental delays.

This proposal is significant because children with special needs are deserving of evidence upon which to base treatment decision-making, but remain under-represented in the medical literature and are often not studied. This research is designed to meet the criteria for the National Institutes of Health road map because it will generate this type of objective evidence that can directly improve patient care.

DETAILED DESCRIPTION:
This will be a prospective, randomized clinical trial. Deaf children (and their parent or guardians) who meet the criteria for developmental delays (as well as the other inclusion and exclusion criteria) will be randomly assigned to receive either hearing aids (group 1) or a cochlear implant (group 2) and followed longitudinally for two years. If one intervention provides improved development and quality of life over the other, this study will provide essential evidence to support clinical decision-making in this population. Children with normal cognition undergoing cochlear implantation will be studied as a control cohort (group 3) in order to demonstrate to what extent the gains after cochlear implantation in children with developmental delays parallel the gains seen in children without developmental delays. There is no placebo group.

Specific aim 1: We will compare the changes in development between the groups. If our hypothesis is true, auditory, linguistic, and cognitive development should demonstrate more improvement in deaf children with developmental delays treated with cochlear implantation compared to those treated with hearing aids.

Specific aim 2: We will compare the changes in quality of life between the groups. If our hypothesis is true, quality of life should demonstrate more improvement in patients treated with cochlear implantation compared to those treated with hearing aids.

Screening will be performed by the Principal Investigator (PI), his collaborators, and his research staff at the Children's Hearing Center at Lucile Packard Children's Hospital (LPCH).

In order to minimize investigator selection bias and in an attempt to produce study groups that are comparable, this is a randomized study. Randomization does not guarantee comparable study groups, particularly in a small trial like this. In order to improve the odds of achieving comparable study groups, we have elected to stratify the randomization process by age. Also, a block randomization process will be used. Lastly, we will compare the groups at the end of the study by looking at their baseline assessment data and stratifying the analysis.

Thus, patients with developmental delays will be randomized into one of two groups after the baseline assessment. This randomization will occur through a specific process in order to assure it is unbiased.

Outcome variables: Four general outcomes will be measured at baseline, one year after the intervention, and two years after the intervention. The first three reflect measures of development (auditory, linguistic, and cognitive; specific aim 1) and the last one is quality of life (specific aim 2).

All data collection will be performed during routine clinic appointments and will not require any special appointments.

All tests will be administered in either English or Spanish, depending on the patient's or their parent's primary language. We have bilingual audiology, speech pathology, and psychology personnel in our center specifically for this purpose. For self-report questionnaires, a Spanish-interpreter provided by the hospital will be used to translate the written materials if a Spanish version of the test is not available. If a parent is not able to read the questionnaire (it is at a 5th grade level), it will be read to them by the testing personnel.

1. Auditory development will be assessed by our cochlear implant audiologists using two different techniques. Behavioral thresholds to speech will be assessed according to standard clinical audiological guidelines. While children hearing through only one cochlear implant cannot localize the sound (two ears are required for this), they will typically demonstrate a behavioral response that indicates cortical perception of the sound. Thus, this data will provide information regarding the ability of the child to hear a sound and then generate a change in behavior. As well, auditory-evoked brainstem response (ABR) or electrically-evoked compound action potential (eCAP) thresholds will be measured in patients wearing their hearing aids or cochlear implant, respectively. These data will also be collected according to standard clinical guidelines.
2. Linguistic development will be assessed by standardized speech and language testing as well as by Systematic Analysis of Language Transcripts (SALT) coding. The standardized tests include the Preschool Language Scale (PLS) and the Peabody Picture Vocabulary Test (PPVT). All testing will be performed by our cochlear implant speech pathologists according to standard clinical guidelines and we already routinely conduct the PLS and PPVT in our clinic. The PLS is used in patients with minimal vocabulary, typically young children, and has been validated from birth to 6 years, 11 months of age. In contrast, the PPVT is more useful in older children who have more vocabulary. It has been validated for children older than 2 years, 6 months of age.

   Another way we propose to study language is through the use of language transcript (SALT) coding. One benefit of this technique is that it permits the test to be adapted to each child's abilities. Thus, there will be follow-up speech and language data on every patient. Importantly, this technique has been used previously to assess the effect of mild-moderate hearing loss and deafness on language development. We will videotape the 30 minute session of the child with one of our speech therapists. This will be performed within a speech therapy room designed for videotaping pediatric patients. The session will be organized by the speech therapist to showcase the child's language abilities according to standard clinical guidelines. These will include the administration of vocabulary tests and either a narrative sample or a conversation and expository sample. The videotape will be coded with no patient identifiers and sent to a collaborator with expertise in infant and child language development who will perform an independent analysis of the tape using SALT coding. The measures that will be will be coded include the Number of Different Words (NDW), Total Number of words (TNW), Mean Length of Utterance (MLU), and nonverbal indicators of comprehension (e.g., via pointing and eyegaze). SALT coding of the videotapes will assess both verbal and non-verbal communication.
3. Cognitive level will be assessed via standardized testing. The Mullen Scales of Early Learning (MSEL) (Pearson, Bloomington, MN) is an objective measure designed for young children to estimate intelligence. The age range for the Mullen is birth to 5 years, 8 months, though it also can be used in older children with significant cognitive impairment such as those included in this study. Items administered for this test load onto 5 different domains (Visual Reception, Gross Motor, Fine Motor, Expressive Language, and Receptive Language). Because verbal and nonverbal domains are assessed separately, this measure is particularly useful in the assessment of children who have suspected language delays and/or hearing loss. We will perform the complete test and analyze the change in each domain (i.e. measured before and after the intervention). The raw scores will be used in order to have the most sensitivity in detecting changes in patients with MR who otherwise would tend to be on the low end of the percentile range. The Vineland Adaptive Behavior Scales (VABS) (Pearson, Bloomington, MN) provides a measure of a child's adaptive functioning. This describes the child's ability to cope and function effectively within their environment. This measure is a structured parent interview and can be performed with caregivers of children from birth to adulthood. In its entirety, the measure provides information regarding a child's functioning across several domains including Communication, Socialization, Motor Skills, and Daily Living Skills. We will perform the complete test and analyze the change in each subscore (i.e. measured before and after the intervention). It is important to note that these are psychological tests that have to be given by a highly-trained pediatric psychologist in the proper environment. The rationale for this precaution is to minimize investigator bias. The neurocognitive data will be collected during a single 3-4 hour visit with our psychologist, who also measured these variables prior to the intervention as part of the Baseline Assessment. Because this testing will always take place by the Psychology Service and in all likelihood by the same examiner, variability will be minimized.
4. Quality of life will be assessed using three standardized techniques. The Parenting Stress Index (PSI) identifies factors increasing the stress in the child-parent system according to parental perception. We have substantial experience using this test measure and have used it with our cochlear implant patients for the last several years. The parental responses are scored and interpreted by the psychologist. The CARE-Index will also be measured with the help of a consultant who originally developed the CARE-Index and has tremendous experience with it. This involves videotaping and analyzing a 3-5 minute "free play" interaction between mother and child. The recording is later coded for maternal attentiveness, infant responsiveness and dyadic interactions using a 14-point sensitivity scale in the CARE-Index.

Intervention:

The intervention for study participants will be performed by dedicated cochlear implant audiologists that will do the cochlear implant or hearing aid programming for this trial. These are highly-trained pediatric audiologists skilled in managing children with complex and severe hearing losses. Thus, the quality of the intervention will be of the highest level, whether it is a cochlear implant or hearing aids.

Patients in group 1 will be fit with bilateral hearing aids. These will be programmed individually for the severity and frequency distribution of hearing loss. The type of hearing aids used will be fit in the most appropriate fashion according to standard audiometric criteria and our clinic norms. Patients in groups 2 and 3 will undergo cochlear implantation. According to Food and Drug Administration guidelines, this can only occur after they reach 12 months of age, unless an extenuating situation exists. As well, all appropriate vaccinations will be in place prior to the surgery, per the guidelines of the Centers for Disease Control (CDC).

Initially, we will only implant one ear. This is the current standard of care and is all that many insurance companies will pay for. The choice of ear will be made on an individual basis, as determined per the routine of the cochlear implant team. This choice depends on the anatomy of the inner ear or auditory nerve and the level of residual hearing in the ears. As well, other factors such as the handedness of the child, the tendency of the child to rest their head on one side or the other, or parental desires also occasionally play into this decision. If the family desires to have a second implant placed in the contralateral ear, we will work with them and their insurance company to try and arrange this.

Patients in all three groups will require frequent follow-up visits to the audiology clinic for device programming. Typically, these visits are more frequent for those patients with a cochlear implant than those with hearing aids, but not always. The schedule for these appointments is made on an individual basis because some children need more frequent changes in device programming than others. If hearing aid molds need to be polished or re-made as the child grows, this will be performed per clinic routine. If cochlear implant software or hardware needs to be updated as new technology emerges, this too will occur per clinic routine. Thus, all patients will be receiving the highest level of care according to current standards. Lost or damaged equipment will be replaced.

As well, patients in all three groups will undergo thorough counseling about hearing loss,and communication strategies. Contact with the child's teachers, therapists, and caregivers will be made in an effort to organize a comprehensive strategy of regular communication therapy. As is our routine, every patient will be offered the opportunity to have supplementary weekly auditory therapy sessions with one of the speech pathologists that are part of our cochlear implant team or through one of our satellite speech pathology clinics. Our speech pathologists can provide auditory-verbal therapy (AVT), although they typically modify the therapy structure to meet the needs of the individual child. Just as with the audiology services, speech pathology services will be of the highest level and quality for children in all groups. However, it should be noted that many families chose not to obtain speech therapy services through our program. Instead, as a matter of convenience, most families choose to have therapy only in their home through free/low cost Early Childhood Intervention (ECI) services or their local school district.

The amount of time the hearing aids or cochlear implant are used and the amount and quality of therapy will be assessed by regular phone calls. Every three months the study coordinator will call the parents/caregiver and ask four questions:

* Have there been any complications of the hearing aids or cochlear implant in the last three months (i.e. ear infections, ear drainage, meningitis), and if so, what therapy was needed for the complication?
* How many hours per day are the hearing aids or cochlear implant are left on the child?
* How many hours per week is the child of communication therapy (defined as auditory, speech, and language therapies) is the child receiving?
* How many hours per week of non-communication therapy (defined as physical, occupational, and cognitive therapies) is the child receiving?

These data will be recorded in the database. The reasons for asking these questions are to identify adverse events related to the interventions and to help identify reasons why one intervention may work better or worse than the other. For example, decreased benefit might be expected if a child treated with hearing aids continuously gets chronic ear drainage that plugs the hearing aids so badly they have to be left off most of the time or if a child treated with a cochlear implant gets meningitis. Alternatively, if receiving a cochlear implant increases the enthusiasm of the parents and they participate in more therapy, there may be increased benefit.

We will also be asking participants if they are willing to be contacted regarding future research studies that may be of interest to them.

ELIGIBILITY:
Inclusion Criteria:

Meet audiometric criteria for cochlear implantation

Age <3 by the time of initiation of treatment

Ability to return for follow-up evaluations at the one and two year time points

Exclusion Criteria:

Evidence of a progressive deteriorating medical condition that may lead to child's death during the time frame of the study

Medical contraindication to cochlear implantation

Significant visual loss

Autism spectrum disorder

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 303 (Actual)
Dates: Start 2009-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
auditory development | two years
Linguistic development | 2 years
Cognitive development | 2 years

SECONDARY OUTCOMES:
Quality of life | two years

CONTACTS AND LOCATIONS:
Overall Officials: John Oghalai, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Sevy AB, Bortfeld H, Huppert TJ, Beauchamp MS, Tonini RE, Oghalai JS. Neuroimaging with near-infrared spectroscopy demonstrates speech-evoked activity in the auditory cortex of deaf children following cochlear implantation. Hear Res. 2010 Dec 1;270(1-2):39-47. doi: 10.1016/j.heares.2010.09.010. Epub 2010 Oct 1. PMID 20888894
- [Background] Lin JW, Mody A, Tonini R, Emery C, Haymond J, Vrabec JT, Oghalai JS. Characteristics of malfunctioning channels in pediatric cochlear implants. Laryngoscope. 2010 Feb;120(2):399-404. doi: 10.1002/lary.20668. PMID 19950369
- [Background] Katzenstein JM, Oghalai JS, Tonini R, Baker D, Haymond J, Caudle SE. Neurocognitive functioning of a child with partial trisomy 6 and monosomy 21. Neurocase. 2009;15(2):97-100. doi: 10.1080/13554790802631910. Epub 2009 Jan 26. PMID 19172430
- [Background] Cristobal R, Oghalai JS. Hearing loss in children with very low birth weight: current review of epidemiology and pathophysiology. Arch Dis Child Fetal Neonatal Ed. 2008 Nov;93(6):F462-8. doi: 10.1136/adc.2007.124214. PMID 18941031
- [Background] Oghalai JS, Tonini R, Rasmus J, Emery C, Manolidis S, Vrabec JT, Haymond J. Intra-operative monitoring of cochlear function during cochlear implantation. Cochlear Implants Int. 2009 Mar;10(1):1-18. doi: 10.1002/cii.372. PMID 18937280
- [Background] Pierson SK, Caudle SE, Krull KR, Haymond J, Tonini R, Oghalai JS. Cognition in children with sensorineural hearing loss: etiologic considerations. Laryngoscope. 2007 Sep;117(9):1661-5. doi: 10.1097/MLG.0b013e3180ca7834. PMID 17690618
- [Background] Kushalnagar P, Krull K, Hannay J, Mehta P, Caudle S, Oghalai J. Intelligence, parental depression, and behavior adaptability in deaf children being considered for cochlear implantation. J Deaf Stud Deaf Educ. 2007 Summer;12(3):335-49. doi: 10.1093/deafed/enm006. Epub 2007 Apr 21. PMID 17449899
- [Background] Choi CH, Oghalai JS. Predicting the effect of post-implant cochlear fibrosis on residual hearing. Hear Res. 2005 Jul;205(1-2):193-200. doi: 10.1016/j.heares.2005.03.018. PMID 15953528
- [Background] Oghalai JS, Chen L, Brennan ML, Tonini R, Manolidis S. Neonatal hearing loss in the indigent. Laryngoscope. 2002 Feb;112(2):281-6. doi: 10.1097/00005537-200202000-00015. PMID 11889384
- [Derived] Oghalai JS, Bortfeld H, Feldman HM, Chimalakonda N, Emery C, Choi JS, Zhou S. Cochlear Implants for Deaf Children With Early Developmental Impairment. Pediatrics. 2022 Jun 1;149(6):e2021055459. doi: 10.1542/peds.2021-055459. PMID 35607935